CLINICAL TRIAL: NCT00462462
Title: Systemic and Local Diffusion of Ethanol After Administration of Ethanol 96% Formulated in a Gel and Ethanol 98% Solution by the Percutaneous Route, in Patients With Congenital Venous Malformations:Pharmacokinetic, Pharmacodynamic and Clinical Study.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orfagen (Industry)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: L00122 GI 201 (ORF)
Record Dates: First submitted 2007-04-16; First posted 2007-04-19 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Congenital Venous Malformation
MeSH Terms: interventions — Ethanol; Gels; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ethanol gel
  Interventions: Drug: Ethanol 96% Gel
- 2 (Active Comparator): Ethanol solution
  Interventions: Drug: Ethanol 98% Solution

INTERVENTIONS:
Drug: Ethanol 96% Gel
  Arms: 1
Drug: Ethanol 98% Solution
  Arms: 2

SUMMARY:
Absolute ethanol has been used "off-label" as an unmodified formulation (solution) in Congenital Venous Malformations (CVM). Despite its effectiveness, absolute ethanol appears difficult to handle because of its high diffusion capacity outside the CVM and in the blood circulation. A less diffusible ethanol-based product (ethanol gel) has been developed in order to minimize systemic and local diffusion capacities of ethanol. Therefore, the pharmacokinetic parameters and their clinical and paraclinical outcomes between ethanol gel 96% and absolute ethanol need to be carried out.

FDA Office of Orphan Products Development (FDA OOPD) : Funding source.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, of at least 12 years of age,
* For women of childbearing potential, negative pregnancy test at baseline,
* Patients with one clinically and radiologically (MRI) documented lesion diagnosed as CVM (pure or predominant),
* Patients for which an embolosclerotherapy by the percutaneous route is indicated as first line therapy of the test lesion, or for which previous treatments (i.e. surgery, embolosclerotherapy, laser) have been unsuccessful or insufficient,
* Patients with CVM lesional size of at least 12 cm3 (maximum craniocaudal dimension X mean dimension of 3 transverse equispaced measurements X mean dimension of 3 deepness equispaced measurements dimension) at MRI,
* Patients with focal or multifocal CVM lesion, i.e. with one or several well-interconnecting venous spaces and well-defined margins,
* Patients or parents able to follow study instructions and attend study visits,
* Written informed consent from the patients or parents.

Exclusion criteria:

* Patients under 12 years of age,
* Pregnant women, nursing mothers and women of childbearing potential with no reliable contraception from more than 2 months,
* Women of childbearing potential with a positive pregnancy test at baseline,
* Patients with CVM of non venous predominance,
* Patients with CVM that are not reachable by the percutaneous route,
* Patients with extensive superficial skin CVM (i.e. with high risk of skin necrosis),
* Patients with a test lesion adjacent to major nerves (e.g. facial nerve in the parotid region, intramuscular regions adjacent to major nerves),
* Patients with facial CVM or bone involvement,
* Patients with small CVM lesion (<12 cm3 at MRI),
* Patients requiring more than 1 ml/Kg body weight (b.w.) in USA or more than 0.5 ml/Kg b.w. in France, or more than 30 mL of absolute ethanol to infuse,
* Patients with a known allergy to one of the components of the test products,
* Patients with a suspected allergy to iodinate.ed products,
* Patients with abnormal clotting parameters (platelets, partial thromboplastin, prothrombin time),
* Patients with an active inflammatory episode of the test lesion (i.e. acute or subacute swelling of the test lesion),
* Patients with complex malformations (e.g. Klippel-Trenaunay syndrome, Blue Rubber Bled Nevus syndrome, Muco-cutaneous familial venous malformations, Mafucci's syndrome),
* Patients in which a surgery, laser therapy or embolosclerotherapy of the test lesion has been performed within the last 12 weeks prior to study entry,
* Asthmatic patients who require daily medications,
* Patients with a non treated or non stabilized cardiac disease,
* Patients with a suspected right-left shunt,
* Patients with an intercurrent condition or a concomitant treatment which may interfere with a good conduct or the evaluation parameters of the study,
* Patients who participated in a study within the 12 weeks prior to study entry,
* Patients or parents who are not able or willing to follow the study instructions,
* Patients or parents who refuse to give written informed consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PATRICK DUPUY, MD, Study Director — ORFAGEN LABORATORIES (France); SALLY E MITCHELL, MD, Principal Investigator — Johns Hopkins Medical Institution (Baltimore, USA); Denis HERBRETEAU, MD, Principal Investigator — Hôpital Bretonneau (Tours, France)
Locations (2):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States
- Hôpital Bretonneau Service de neuroradiologie, Tours, France

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 32 patients were enrolled in the study, but 31 received the study product (1 patient not treated; inclusion mistake).
Groups:
- L0122 Gel Group: Patients who received one intralesional administration of L0122 gel
- Absolute Ethanol Group: Patients who received one intralesional administration of Absolute Ethanol
Period: Overall Study
Arm/Group | L0122 Gel Group | Absolute Ethanol Group
Started | 17 | 14
Completed | 17 | 13
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of the patients who received the study product (L0122 gel or Absolute Ethanol), whichever the amount of product was infused . 32 patients were enrolled in the study, but 31 received the study product (1 patient not treated; inclusion mistake).
Groups:
- Total: Total of all reporting groups
Arm/Group | L0122 Gel Group | Absolute Ethanol Group | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 2 | 7
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  France | 8 | 7 | 15
  United States | 9 | 7 | 16
Lesional volume [Mean (Standard Deviation); unit: cm3] | 82.712 (156.316) | 561.472 (1147.306) | 298.926 (801.306)

OUTCOME MEASURES:

1. Primary Outcome: Systemic Exposure to Ethanol With the Two Test Products: Determination of the Maximum Plasma Concentration (Cmax)
Description: Blood samples were performed, just before infusion, then 5 min, 10 min, 20 min, 40 min, 60 min, 90 min, and 120 min after infusion at the first site, then every 60 min onwards until ethanol levels are found under the detection limit. Cmax was estimated directly from experimental data. If all the ethanol concentrations of a patient was below the limit of quantification of the laboratory (LOQ), Cmax was reported as LOQ/2 for this patient.
Time Frame: Baseline visit (just before and during test product infusion procedure)
Measure: Mean (Full Range); unit: g/L
Groups:
- L0122 Gel Group: Patients who received one intralesional administration of L0122 gel and who had blood samples just before and during infusion procedure.
- Absolute Ethanol Group: Patients who received one intralesional administration of Absolute Ethanol and who had blood samples just before and during infusion procedure (one patient who received Absolute Ethanol was not sampled during infusion procedure).
Arm/Group | L0122 Gel Group | Absolute Ethanol Group
Number analyzed (Participants) | 17 | 13
g/L | 0.0604 [0.015 to 0.4] | 0.202 [0.05 to 0.940]

2. Secondary Outcome: Systemic (Cardiopulmonary, Hematological, Metabolic) and Local Outcome of the Two Test Products.
Time Frame: Study end
Reporting Status: Not Posted

3. Secondary Outcome: Change in Volume of Congenital Venous Malformation (CVM) From Screening to Study End (Day 112 Visit).
Time Frame: Screening and study end (Day 112)
Measure: Mean (Standard Deviation); unit: cm3
Groups:
- L0122 Gel Group: Patients who received one intralesional administration of L0122 gel and for whom lesional volume measurements were available at screening and at study end
- Absolute Ethanol Group: Patients who received one intralesional administration of Absolute Ethanol and for whom lesional volume measurements were available at screening and at study end
Arm/Group | L0122 Gel Group | Absolute Ethanol Group
Number analyzed (Participants) | 17 | 13
cm3 | -10.328 (36.667) | -126.944 (367.229)

4. Secondary Outcome: Patient Benefit
Time Frame: study end
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | L0122 Gel Group | Absolute Ethanol Group
Serious Adverse Events (participants affected / at risk) | 2/17 | 4/14
Other Adverse Events (participants affected / at risk) | 12/17 | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | L0122 Gel Group (N=17) | Absolute Ethanol Group (N=14)
Blood ethanol increased (Investigations) | 0 | 3
Arteriovenous malformation (Congenital, familial and genetic disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | L0122 Gel Group (N=17) | Absolute Ethanol Group (N=14)
Injection site paraesthesia (General disorders) | 3 | 0
Pain (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Injection site discolouration (General disorders) | 1 | 0
Injection site extravasation (General disorders) | 1 | 0
Injection site thrombosis (General disorders) | 1 | 0
Complication of device insertion (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Injection site ulcer (General disorders) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 2 | 4
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 0
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 2 | 4
Coagulopathy (Blood and lymphatic system disorders) | 1 | 5
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Fibrin degradation products increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Haemoglobinuria (Renal and urinary disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days